CLINICAL TRIAL: NCT00212745
Title: Nonrandomized Pilot Trial of the Andrews/Reiter Behavioral Treatment for Epilepsy
Brief Title: Pilot Trial of a Behavioral Treatment for Epilepsy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRF #0425; MRF #0425
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Epilepsies, Partial
Keywords: Behavior Therapy; Relaxation Techniques
MeSH Terms: conditions — Epilepsies, Partial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (No Intervention): Receives only EEG and questionnaire testing, no behavioral intervention or meditative relaxation
- 1 (Experimental): Andrews/Reiter behavioral treatment for epilepsy and EEG and questionnaire testing
  Interventions: Behavioral: Andrews/Reiter behavioral treatment for epilepsy

INTERVENTIONS:
Behavioral: Andrews/Reiter behavioral treatment for epilepsy — The behavioral intervention in this study uses lifestyle counseling to avoid triggers for seizures and strategies to stop beginning seizures. Participants are taught to practice meditative relaxation exercises.
  Arms: 1

SUMMARY:
The purpose of this research study is to see if a behavioral program which includes a relaxation technique and lifestyle changes can improve seizure control and well-being in epilepsy patients.

DETAILED DESCRIPTION:
The behavioral treatment approach studied aims to help epilepsy patients discover which circumstances and behaviors trigger their seizures. The most common seizure precipitants are irregularities of sleep, sensory triggers such as flashing lights and emotional stress. Patients will learn how to avoid seizure precipitants and how to stop seizures in their first beginnings. Study participants will continue their prior medications.

ELIGIBILITY:
Inclusion Criteria:

* Age 16-50 years.
* Reliable diagnosis of partial epilepsy, including simple or complex partial or secondarily generalized tonic-clonic seizures.
* Average seizure frequency of at least one partial seizure per month for at least one year.
* Willing not to begin another new treatment other than anticonvulsants (acupuncture, botanicals or other mind-body interventions, ketogenic diet, vagus nerve stimulator, or epilepsy surgery) while enrolled in the study.

Exclusion Criteria:

* Unreliable history of seizure semiology.
* Average seizure frequency less than one seizure per month.
* Patients in whom it is anticipated that current standard of care would mandate a change in their conventional epilepsy treatment during the time period of the study will be excluded.
* Patients taking more than 2 anticonvulsant medications will be excluded.
* Patients with serious other medical problems, such as brain tumors, cancer, stroke, significant heart disease or psychiatric disorders will be excluded.
* Patients with a high likelihood of psychogenic or nonepileptic seizures will be excluded.
* Patients with progressive epilepsy syndromes, neurodegenerative disorders or significant mental retardation will be excluded.

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2004-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Seizure frequency | At enrollment, end of 2-3 month baseline, after 6 months of treatment, and 6 months after end of treatment.

SECONDARY OUTCOMES:
Epileptiform EEG changes | At enrollment, end of 2-3 month baseline, after 6 months of treatment, and 6 months after end of treatment.
Heartrate variability | At enrollment, end of 2-3 month baseline, after 6 months of treatment, and 6 months after end of treatment.
Salivary cortisol | At enrollment, end of 2-3 month baseline, after 6 months of treatment, and 6 months after end of treatment.
Questionnaires on stress, emotional well-being, self-efficacy, sleepiness and quality of life | At enrollment, end of 2-3 month baseline, after 6 months of treatment, and 6 months after end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Siegward M Elsas, M.D., Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States